CLINICAL TRIAL: NCT05146271
Title: Change in Quality of Life After Full Mouth Rehabilitation Under General Anesthesia in a Group of Egyptian Children With Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mmohamed ramadan mohamed ahmed, Cairo university, Cairo University
Other Study IDs: Change in quality of life
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Complete mouth rehabilitation under general anesthesia in a group of Egyptian children with Down syndrome — Complete mouth rehabilitation under general anesthesia in a group of Egyptian children with Down syndrome

SUMMARY:
To assess oral health related quality of life (OHRQOL) after full mouth rehabilitation under GA in a group of Egyptian children with down syndrome .

DETAILED DESCRIPTION:
Dental treatment under GA provides a safe approach and has significant positive effects on quality of life for children with down syndrome who cannot accept normal treatment. Oral health related quality of life is measured in relation to how the mouth and teeth affect physical, psychological and social well-being and daily activities such as eating, chewing, swallowing, speaking, playing, learning, happiness, embarrassment, and social interactions (Jabarifar et al., 2009). Jankauskiene et al., 2010 conducted a systematic review concluded that "Oral rehabilitation under GA results in immediate improvement of the children's oral health and physical, emotional and social quality of life. It also has a positive impact on the family". Dental caries is a common condition amongst young children which negatively impacts on their quality of life. children with down syndrome who have an increased risk of developing caries due to various reasons: limited oral healthcare, difficultty in dental services,un stable diet, the high sugar contents in their medications and low salivary secretion(Peerbhay & Titinchi, 2014).

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria Age range 1 to 15 years. Diagnosed with down syndrome Should have a minimum of 12 primary or permanent teeth, or a mixture that had not been treated within the past 12 months.

Exclusion Criteria Participation in any other concurrent clinical trials. The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.

Children whose parents had no home or mobile phone to enable post-operative contact.

Parent that will not sign the consent.

Exclusion Criteria:

* Inclusion Criteria Age range 3 to 14 years. Diagnosed with down syndrome Should have a minimum of 12 primary or permanent teeth, or a mixture that had not been treated within the past 12 months.

Exclusion Criteria Participation in any other concurrent clinical trials. The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.

Children whose parents had no home or mobile phone to enable post-operative contact.

Parent that will not sign the consent.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group of Egyptian Children with Down Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
assess oral health related quality of life (OHRQOL) after full mouth rehabilitation under GA in a group of Egyptian children with down syndrome . | Baseline
  assess oral health related quality of life (OHRQOL) after full mouth rehabilitation under GA in a group of Egyptian children with down syndrome .

SECONDARY OUTCOMES:
Change in family conflict scale | Baseline
  Change in family conflict